CLINICAL TRIAL: NCT06792214
Title: Antiviral Strategies in the Prevention of Long-term Cardiovascular Outcomes Following COVID-19: The paxloviD/Remdesivir Effectiveness For the prEvention of loNg coviD (DEFEND) Clinical Trial
Brief Title: Antiviral Strategies in the Prevention of Long-term Cardiovascular Outcomes Following COVID-19: The paxloviD/Remdesivir Effectiveness For the prEvention of loNg coviD Clinical Trial
Acronym: DEFEND
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: Unity Health Toronto (Other); Kingston Health Sciences Centre (Other); Niagara Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UTN: U1111-1311-3673; 202309PPE (Other Grant/Funding Number: CIHR); 185352 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2024-12-23; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-12

CONDITIONS: SARS CoV-2 Post-Acute Sequelae
Keywords: SARS CoV-2; long covid
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — nirmatrelvir and ritonavir drug combination; remdesivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Paxlovid (Experimental): Paxlovid vs. placebo
  Interventions: Drug: Nirmatrelvir/ritonavir
- Veklury (Experimental): Veklury vs. placebo
  Interventions: Drug: Remdesivir

INTERVENTIONS:
Drug: Nirmatrelvir/ritonavir — Paxlovid PO BID for 5 days + standard of care
  Other Names: Paxlovid
  Arms: Paxlovid
Drug: Remdesivir — Veklury IV daily for 5 days + standard of care
  Other Names: Veklury
  Arms: Veklury

SUMMARY:
The DEFEND trial will be the world's first clinical trial to study the effectiveness of Paxlovid or Veklury in the prevention of cardiovascular post-acute sequelae of SARS-CoV-2 among hospitalized adults. Additionally, this pilot study will inform the design and conduct of a future full-scale multi-centre trial by testing the feasibility and accuracy of this study design.

DETAILED DESCRIPTION:
The overall goal of the DEFEND clinical trial is to study the effectiveness of Paxlovid or Veklury in preventing cardiovascular post-acute among adults who test positive for SARS-CoV-2 at admission to hospital. The pilot trial will inform the design and conduct of a future full-scale multicentre trial by estimating the feasible recruitment rate. Our secondary aim is to validate the accuracy of hospital-based outcome measures in administrative data, and to determine the event rate of a composite of any of 4 newly developed or worsening stroke, heart failure, venous thromboembolism, diabetes or death within 1 year. The DEFEND trial will be a pragmatic, multicentre, registry-based, double-blind, two-arm, randomized placebo-controlled internal pilot trial. If no major protocol changes are required, the data obtained from the pilot will be included in the future large trial; if major protocol changes are required, the results from the pilot trial will still be published and will be useful to inform future research in this area. The approach is pragmatic to include as many participants as possible that could benefit from treatment with Paxlovid or Veklury using broad eligibility criteria for enrolment and reflecting the real world practice of treating physicians. The DEFEND trial will enrol participants aged ≥18 who have a positive polymerase chain reaction test for SARS-CoV-2 at admission to 4 hospitals in Ontario. If they meet the inclusion/exclusion criteria they will be randomized to either the experimental or control arm of the trial. Those in the experimental arm will receive either Paxlovid orally twice daily for 5 days or Veklury intravenously once daily for 5 days (as well as standard of care). Those in the control arm will receive the placebo at the same schedule and frequency for 5 days (as well as standard of care). Randomization will be at a 1:1 allocation, stratified by hospital. The DEFEND trial seeks to enrol 118 participants at 4 committed pilot trial sites that are representative of acute care hospitals across Ontario over a 12 month period. This will be followed by a 12 month follow-up period. The DEFEND trial will be the world's first clinical trial to study the effectiveness of Paxlovid or Veklury in the prevention of cardiovascular post-acute sequelae of SARS-CoV-2 among hospitalized adults.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Positive PCR test for SARS-CoV-2 within 5 days of admission to hospital
* Normoxic (not receiving supplemental oxygen)
* Able to provide informed written consent (or, if patient is unable, have substitute decision maker available)

Exclusion Criteria:

* Absolute contraindications to Paxlovid or Veklury (any of the following): Severe allergy to Paxlovid or Veklury (e.g. anaphylaxis), co-administration with drugs highly dependent on CYP3A for clearance, co-administration with potent CYP3A inducers
* Exposure to Paxlovid or Veklury within previous 14 days;
* Receiving supplemental oxygen;
* Known positive SARS-CoV-2 PCR or rapid antigen test 5-90 days prior to admission;
* Limited life expectancy estimated to be ≤3 months;
* Pregnant and breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2025-01-03 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | From participant screening to enrolment
  Recruitment rate, defined as the proportion of eligible people who consent and are randomized into the pilot trial, which will inform the feasibility of a full scale trial.
Post-acute sequelae of COVID-19 (PASC) | From enrolment to end of follow up at 1 year
  Event rate of PASC at 1 year (specifically newly developed or worsening: stroke, heart failure, venous thromboembolism, diabetes or death)

SECONDARY OUTCOMES:
Administrative data validation | From enrolment to end of follow up at 1 year
  Validate the accuracy of using administrative data to collect participant hospital-based outcome measures including:
  1. Adherence to treatment, measured by whether the participant received the study drug or not as documented in the medication administration record.
  2. Use of co-interventions (dexamethasone, tocilizumab/sarilumab, baricitinib) owing to progression of disease severity as measured by spO2 <92%
  3. Time to treatment initiation, as measured by the time between randomization and first treatment dose.
  The validation of administrative data will be assessed by comparing concordance between manually collected data by research coordinators entered into REDCap and the GEMINI administrative database for the measures described above.
Reinfection, ICU admission, and drug safety | From enrolment to 90 days after initial PCR positive test for COVID-19
  Any of the following treatment related adverse events as assessed with the CTCAE v6.0:
  1. Number and percentage of participants hospitalized with SARS-CoV-2 reinfection within 90 days following initial PCR positive test for COVID-19;
  2. Number and percentage of participants admitted to ICU during initial hospitalization;
  3. Number and percentage of participants experiencing any one of the following adverse study drug effects including dysgeusia, vomiting, or diarrhea as identified by their most responsible physician

CONTACTS AND LOCATIONS:
Locations (4):
- Canada (4):
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Niagara Health System, St. Catharines, Ontario
  - Mount Sinai Hospital, Sinai Health System, Toronto, Ontario
  - St. Joseph's Health Centre, Unity Health Toronto, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Undecided